CLINICAL TRIAL: NCT00458822
Title: Risk-Adapted Intravenous Melphalan With Stem Cell Transplant and Adjuvant Bortezomib and Dexamethasone for Recently Diagnosed Untreated Patients With Systemic Light-Chain (AL) Amyloidosis
Brief Title: Melphalan and Autologous Stem Cell Transplant Followed By Bortezomib and Dexamethasone in Treating Patients With Previously Untreated Systemic Amyloidosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-006; MSKCC-07006
Record Dates: First submitted 2007-04-09; First posted 2007-04-11 (Estimated); Results first posted 2016-08-10 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-06

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: primary systemic amyloidosis
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell; Immunoglobulin Light-chain Amyloidosis | interventions — Bortezomib; Dexamethasone

ARMS (1):
- All Patients (Experimental): All patients treated with Melphalan with Stem Cell Transplant and Adjuvant Bortezomib and Dexamethasone for Recently Diagnosed Untreated Patients with Systemic Light-Chain (AL) Amyloidosis
  Interventions: Drug: bortezomib; Drug: dexamethasone

INTERVENTIONS:
Drug: bortezomib — Given IV
Drug: dexamethasone — Given orally

SUMMARY:
The purpose of this study in patients needing treatment for AL amyloidosis is to see how well treatment with IV melphalan works and then, if some clonal plasma cells are still present about 2 to 3 months after melphalan treatment, to see how well treatment with bortezomib and dexamethasone works to reduce the rest of the clonal plasma cell disease.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed amyloidosis

  * Diagnosed within the past 12 months
  * Clonal plasma cell disorder, as demonstrated by any of the following:

    * Presence of M-protein in serum and/or urine by immunofixation and/or serum free light chain assay
    * Clonal population of plasma cells in the bone marrow based on kappa/lambda staining of a marrow biopsy
* Negative genetic testing for hereditary forms of amyloidosis
* No amyloid-specific syndrome (e.g., carpal tunnel syndrome or skin purpura) as the only evidence of disease

  * Vascular amyloidosis only in a bone marrow biopsy specimen or in plasmacytoma is not indicative of systemic amyloidosis
* No advanced cardiac amyloidosis
* Must have symptomatic involvement of no more than 2 of the following visceral organ systems:

  * Kidneys
  * Liver/gastrointestinal
  * Peripheral/autonomic nervous system
  * Heart
* No persistent pleural effusions
* No clinically overt multiple myeloma with > 30% plasma cells in the bone marrow or lytic bone lesions
* Able to undergo autologous stem cell transplantation

PATIENT CHARACTERISTICS:

* SWOG performance status 0-3
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Bilirubin < 2.0 mg/dL
* Creatinine clearance < 51 mL/min allowed
* LVEF > 45% by echocardiogram
* No New York Heart Association class III-IV congestive heart failure
* No history of cardiac syncope
* No recurrent symptomatic arrhythmias
* No oxygen-dependent restrictive cardiomyopathy
* No myocardial infarction within the past 6 months
* Pulmonary diffusion capacity > 50% predicted by pulmonary function testing
* No uncontrolled infection
* No other active malignancy, except for any of the following:

  * Adequately treated basal cell or squamous cell skin cancer
  * In situ cervical cancer
  * Adequately treated stage I cancer from which the patient is currently in complete remission
  * Any other cancer from which the patient has been disease-free for 5 years
* No hypersensitivity to bortezomib, boron, or mannitol
* No HIV positivity
* No serious medical or psychiatric illness that would preclude study compliance

PRIOR CONCURRENT THERAPY:

* At least 14 days since prior investigational drugs
* No prior therapy for monoclonal plasma disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather Landau, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Patients
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 40
Age, Continuous [Median (Full Range); unit: years] | 57 [38 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 17

OUTCOME MEASURES:

1. Primary Outcome: Hematologic and Organ Response
Description: patients will be assessed for hematologic response (the response of the clonal plasma cell disease). If the plasma cell disease persists, then they will receive 6 cycles of adjuvant therapy with bortezomib and dexamethasone; patients with peripheral neuropathy will receive dexamethasone alone because of the risk of neuropathy associated with bortezomib. Symptomatic organ involvement with amyloid as defined below. Patients must have symptomatic involvement of no more than 2 of the following 4 visceral organ-systems: kidneys, liver/GI, peripheral/autonomic nervous system, and heart.
Time Frame: 2-3 months post transplant
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 40
participants
  Complete Hematologic Response | 11
  Partial Response | 7
  Stable Disease | 18

ADVERSE EVENTS:
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 20/40
Other Adverse Events (participants affected / at risk) | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=40)
Arthritis (non-septic) (General disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
CNS cerebrovascular ischemia (Nervous system disorders) | 1 (1)
Cardiac Arrhythmia, other (Cardiac disorders) | 1 (1)
Cardiac General, other (Cardiac disorders) | 6 (6)
Coagulation, other (Blood and lymphatic system disorders) | 2 (2)
Conduction Abnormality NOS (General disorders) | 1 (1)
Death not associated with CTCAE term- Death NOS (General disorders) | 3 (3)
Dehydration (Gastrointestinal disorders) | 1 (2)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Febrile neutropenia (General disorders) | 1 (1)
Fever (in the absence of neutropenia) (General disorders) | 1 (1)
Hemorrhage, Upper GI NOS (Gastrointestinal disorders) | 1 (1)
Hemorrhage/Bleeding, other (General disorders) | 1 (1)
Hypotension (Cardiac disorders) | 4 (5)
Hypoxia (General disorders) | 1 (1)
Neutrophil-Pneumonia (lung) (Infections and infestations) | 2 (2)
Neutrophil-Up airway NOS (Infections and infestations) | 1 (1)
Infection, other (Infections and infestations) | 5 (5)
Nausea (Gastrointestinal disorders) | 1 (1)
Ocular/Visual - Other (General disorders) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 4 (4)
Pulm/upper respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 3 (3)
Restrictive cardiomyopathy (Cardiac disorders) | 1 (2)
Sodium, low (hyponatremia) (Metabolism and nutrition disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Syncope (fainting) (Nervous system disorders) | 4 (4)
Thrombosis/thrombus/embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Vasovagal episode (Nervous system disorders) | 2 (2)
Ventricular arrhythmia- Ventricular tachycardia (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=40)
Albumin, low (hypoalbuminemia) (Metabolism and nutrition disorders) | 31
Alkaline phosphatase (Metabolism and nutrition disorders) | 9
ALT, SGPT (Blood and lymphatic system disorders) | 11
AST, SGOT (Blood and lymphatic system disorders) | 6
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 5
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 6
Cholesterol,high(hypercholestremia) (General disorders) | 6
Constipation (Gastrointestinal disorders) | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Creatinine (Metabolism and nutrition disorders) | 22
Cushingoid appearance (General disorders) | 2
Dehydration (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 3
Distension/bloating, abdominal (Gastrointestinal disorders) | 3
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 4
Fatigue (asthenia, lethargy, malaise) (General disorders) | 15
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 27
Glucose, low (hypoglycemia) (Metabolism and nutrition disorders) | 12
Hemoglobin (Blood and lymphatic system disorders) | 37
Infection, other (Infections and infestations) | 2
Prothrombin Time international normalized ratio (Blood and lymphatic system disorders) | 10
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 38
Lipase (General disorders) | 2
Lymphopenia (Blood and lymphatic system disorders) | 39
Magnesium, high (hypermagnesemia) (Metabolism and nutrition disorders) | 5
Magnesium, low (hypomagnesemia) (Metabolism and nutrition disorders) | 2
Nausea (Gastrointestinal disorders) | 4
Neuropathy: sensory (Nervous system disorders) | 10
Neutrophils/granulocytes (Blood and lymphatic system disorders) | 36
Pain - Neuralgia/peripheral nerve (Nervous system disorders) | 7
Phosphate, low (hypophosphatemia) (Metabolism and nutrition disorders) | 18
Platelets (Blood and lymphatic system disorders) | 39
Potassium, high (hyperkalemia) (Metabolism and nutrition disorders) | 9
Potassium, low (hypokalemia) (Metabolism and nutrition disorders) | 14
Pruritus/itching (Skin and subcutaneous tissue disorders) | 2
Partial thromboplastin time (Blood and lymphatic system disorders) | 5
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2
Renal failure (Renal and urinary disorders) | 2
Sodium, low (hyponatremia) (Metabolism and nutrition disorders) | 12
Syncope (fainting) (Nervous system disorders) | 3
Weight gain (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes